CLINICAL TRIAL: NCT00425737
Title: A Study to Assess the Efficacy, Immunogenicity and Safety of Two Doses of Oral Live Attenuated Human Rotavirus (HRV) Vaccine (Rotarix) in Healthy Infants.
Brief Title: Assess Efficacy, Immune Response & Safety of 2 Doses of Oral Live Attenuated HRV Vaccine in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 444563/004
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Rotavirus
Keywords: Oral live attenuated human rotavirus vaccine; Gastroenteritis
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — RIX4414 vaccine

INTERVENTIONS:
Biological: Rotarix

SUMMARY:
To assess the efficacy, immune response and safety of the oral live attenuated HRV vaccine (Rotarix) in healthy infants approximately 2 months of age and previously uninfected with human rotavirus

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 6 and 12 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parents or guardians of the subject.
* Born after a normal gestation period (between 36 and 42 weeks).

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the study vaccine or placebo or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth. (Topical steroids are allowed.)
* Use of antibiotics during the period starting from 7 days before each dose of vaccine(s) and ending 7 days after.
* Any clinically significant history of chronic gastrointestinal disease or other serious medical condition as determined by the investigator.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine.
* Gastroenteritis within 7 days preceding the study vaccine administration (warrants deferral of the vaccination).
* Household contact with an immunosuppressed individual or pregnant woman.
* Abnormal stool pattern.
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period.
* Previous confirmed occurrence of rotavirus gastroenteritis.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 405 (Actual)
Dates: Start 2000-08; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of RV GE

SECONDARY OUTCOMES:
Occurrence of severe RV GE, solicited symptoms (Day 0-14), unsolicited Adverse Events (Day 0-42), Serious Adverse Events (full study), presence of rotavirus antigen in stool samples, immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] De Vos B, Vesikari T, Linhares AC, Salinas B, Perez-Schael I, Ruiz-Palacios GM, Guerrero Mde L, Phua KB, Delem A, Hardt K. A rotavirus vaccine for prophylaxis of infants against rotavirus gastroenteritis. Pediatr Infect Dis J. 2004 Oct;23(10 Suppl):S179-82. doi: 10.1097/01.inf.0000142370.16514.4a. PMID 15502699
- [Background] De Vos B, Han HH, Bouckenooghe A, Debrus S, Gillard P, Ward R, Cheuvart B. Live attenuated human rotavirus vaccine, RIX4414, provides clinical protection in infants against rotavirus strains with and without shared G and P genotypes: integrated analysis of randomized controlled trials. Pediatr Infect Dis J. 2009 Apr;28(4):261-6. doi: 10.1097/INF.0b013e3181907177. PMID 19289978
- [Background] Soriano-Gabarró M et al. (2008) Potential impact of Rotarix according to rotavirus type distribution. Pediatr Infect Dis J. 27(1):28-32.
- [Background] Vesikari T et al. (2003) Efficacy of oral human rotavirus vaccine in infants against acute rotavirus gastroenteritis in the community determined with rotavirus antigen detection by EIA and rotavirus RT-PCR as end points. J Clin Virol. 27(1):8 (Abstract n° 24).
- [Background] Vesikari T, Karvonen A, Puustinen L, Zeng SQ, Szakal ED, Delem A, De Vos B. Efficacy of RIX4414 live attenuated human rotavirus vaccine in Finnish infants. Pediatr Infect Dis J. 2004 Oct;23(10):937-43. doi: 10.1097/01.inf.0000141722.10130.50. PMID 15602194
- [Background] Vesikari T, Karvonen A, Puustinen L, Szakal ED, Zeng SQ, Delem A, De Vos B. A short report on highlights of world-wide development of RIX4414: an European experience. Vaccine. 2006 May 1;24(18):3779. doi: 10.1016/j.vaccine.2005.07.028. Epub 2005 Aug 1. No abstract available. PMID 16581159
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 444563/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 444563/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 444563/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 444563/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 444563/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 444563/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register